CLINICAL TRIAL: NCT05111392
Title: Hydration Dynamics and Influence of Beverage Composition
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Craig A. Horswill, Clinical Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0823; Abbott Nutrition (EAS) (Other Grant/Funding Number: Non-Federal Industry)
Record Dates: First submitted 2021-11-04; First posted 2021-11-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hydration; Fluid Retention; Dehydration
Keywords: Hydration; Deuterium oxide; Plasma osmolality; Sodium; Urine production; Fluid absorption; Euhydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: Mixed model.
Who Masked: Participant
Masking Description: Beverages will have similar color, flavoring, and taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Water
  Interventions: Biological: Placebo
- Oral rehydration solution 1 (Experimental): Beverage with 2.5% glucose with 45 mmol sodium/L.
  Interventions: Biological: Oral Rehydration Solution 1
- Oral rehydration solution 2 (Experimental): Beverage with 1.7% glucose with 60 mmol sodium/L.
  Interventions: Biological: Oral Rehydration Solution 2

INTERVENTIONS:
Biological: Placebo — Ingestion of one (1) liter of beverage with observation for 2 h
  Arms: Placebo
Biological: Oral Rehydration Solution 1 — Ingestion of one (1) liter of beverage with observation for 2 h
  Arms: Oral rehydration solution 1
Biological: Oral Rehydration Solution 2 — Ingestion of one (1) liter of beverage with observation for 2 h
  Arms: Oral rehydration solution 2

SUMMARY:
The study examines interactions between fluid availability in the gut and fluid retention in the body. The relative rate of fluid uptake, the expansion of the plasma volume, and percent of fluid retained by the body will be measured in response to ingestion of beverages of different composition. Healthy, euhydrated adults will be studied. The results will help establish formulations of beverages that sustain if not promote acute euhydration.

DETAILED DESCRIPTION:
Using a randomized order for beverage treatments at three separate trials, subjects will ingest 1 Liter of one of three beverages in 10 minutes: water, a beverage with 2.5% glucose with 45 mmol sodium/L, or a beverage with 1.7% glucose with 60 mmol sodium/L. Before and repeatedly for 2 h after ingestion of the beverage, blood samples will be drawn for assessments of D2O, Hb, Hct, osmolality, sodium, and glucose. The rate of appearance of D2O will be evaluated using the area under the curve, the slope of the appearance, and half time to plateau. Comparisons will be made between beverages for indices of the rate of appearance of D2O, the change in PV over time, and cumulative urine excreted. The cumulative urine produced will be used to calculate a modified BHI for the two glucose-electrolyte beverages and water for comparison with 1.0 (expected for no beverage effect). We hypothesize faster absorption (D2O appearance rate), and better overall hydration (expanded PV and higher modified BHI) will occur for beverages containing glucose and sodium compared to water. Further, we hypothesize that of the electrolyte beverages, the beverage with higher sodium content will promote greater overall hydration (less urine excreted) than the beverage with lower sodium.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of 18.5 to 29.9 kg/m2.
* Be normotensive (<120/80 mm Hg).
* Must be able to speak and read English.
* Be physically active or a regular exerciser but be able to abstain from exercise for 48 h prior to each study trial.
* Fast for at least 8 hours prior to and through the study trial.
* Be able to abstain from alcohol for 48 h prior to each study.
* Be able to abstain from caffeine for 24 h prior to each study.
* If female, must have regular menstrual cycles, that are > 27 days and < 35 days in length.

Exclusion Criteria:

* Under 18 y of age or over 45 y of age.
* Have a BMI <18.5 or >30.
* Being pregnant.
* Lactating.
* Tobacco user.
* Have hypotension or hypertension.
* Have any type of kidney disease or dysfunction.
* Have diabetes.
* Have any type of cardiovascular disease.
* Have been diagnosed with galactosemia.
* Females with irregular menstrual cycles.
* Females with polycystic ovary disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of appearance of deuterium in the plasma for placebo | 2 hours
  Measure the rate of fluid uptake by the gut using appearance of deuterium oxide, or D2O, in the blood after ingesting a fixed volume of placebo.
Rate of appearance of deuterium in the plasma for oral rehydration solution 1. | 2 hours
  Measure the rate of fluid uptake by the gut using appearance of deuterium oxide, or D2O, in the blood after ingesting a fixed volume of placebo.
Rate of appearance of deuterium in the plasma for oral rehydration solution 2. | 2 hours
  Measure the rate of fluid uptake by the gut using appearance of deuterium oxide, or D2O, in the blood after ingesting a fixed volume of placebo.

SECONDARY OUTCOMES:
Fluid retention for placebo | 2 hours
  Measure fluid retention using the difference between ingested volume and cumulative urine excretion as a percentage of the ingested volume.
Fluid retention for oral rehydration solution 1 | 2 hours
  Measure fluid retention using the difference between ingested volume and cumulative urine excretion as a percentage of the ingested volume.
Fluid retention for oral rehydration solution 2 | 2 hours
  Measure fluid retention using the difference between ingested volume and cumulative urine excretion as a percentage of the ingested volume.
Change in plasma volume for placebo | 2 hours
  Increase in plasma volume (water content of the blood) following ingestion of beverage
Change in plasma volume for oral rehydration solution 1 | 2 hours
  Increase in plasma volume (water content of the blood) following ingestion of beverage
Change in plasma volume for oral rehydration solution 2 | 2 hours
  Increase in plasma volume (water content of the blood) following ingestion of beverage

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Horswill, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
If shared, the main outcome variables will be posted.